CLINICAL TRIAL: NCT04560790
Title: CRISPR/Cas9 mRNA Instantaneous Gene Editing Therapy Assisted Corneal Transplantation in the Treatment of Refractory Viral Keratitis
Brief Title: Safety and Efficacy of CRISPR/Cas9 mRNA Instantaneous Gene Editing Therapy to Treat Refractory Viral Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JYMS-CXL#02
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Viral Keratitis; Blindness Eye; Herpes Simplex Virus Infection; Cornea
Keywords: Herpes simplex virus type 1 (HSV-1); CRISPR/Cas9 mRNA; instantaneous gene editing
MeSH Terms: conditions — Blindness; Herpes Simplex; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Single group target value: Since there is no similar products approved on the market and there is no similar comparative treatment methods, the single group target value method is adopted
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BD111 Adults single group Dose (Experimental): Administered by corneal injection surgery. Dosage form:injection solution. Dose:200uL. Frequency of administration: one time injection.
  Interventions: Drug: BD111 Adult single group Dose

INTERVENTIONS:
Drug: BD111 Adult single group Dose — 3-6 Participants will receive a single group dose administered via corneal injection in the study eye.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of a single escalating doses of BD111 CRISPR/Cas9 mRNA Instantaneous Gene Editing Therapy administered via corneal injection in participants with refractory herpetic viral keratitis.

DETAILED DESCRIPTION:
This is an open-label, single ascending dose study of BD111 in adult (ages 18 to 70) participants with refractory herpetic viral keratitis. Approximately 6 participants will be enrolled.BD111 is a novel gene editing product designed to clear Herpes simplex virus type I (HSV-1) that results in herpetic stromal keratitis in both acute and recurrent infection models which is the leading factor for infectious blindness.

The follow-up period was 360 days, and the patients will be followed up 3±1 days, 7±2 days, 30±7 days, 90±14 days, 180±21 days, and 360+31 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients (replase) with refractory keratitis caused by herpes virus type I who has had at least one time failed corneal transplant.

1. Age between 18 to 70 years.
2. No systemic immune eye disease.
3. Good eyelid structure and blink function.
4. Exists the potential of visual recovery by evaluation of ocular structure and function.
5. Patients with refractory keratitis who are repeatedly infected with HSV-1 virus (more than three times per year) and resistant to topical or systemic anti-viral agents, with no response to regular immunosuppressive agents.
6. Patients who are obviously suffering from relapse HSV infections with corneal perforation, requiring corneal transplantation;
7. No history of corneal trauma.
8. Subjects or their legal guardians voluntarily participate in this study, sign informed consent, good compliance and cooperation with follow-up visits.

Exclusion Criteria:

1. Lacrimal coating and blink function loss.
2. Schirmer's test result is less than 2mm for severe dry eye disease.
3. Pregnant and lactating women (pregnancy defined in this study as positive urine pregnancy test).
4. Currently is involved in clinical trials of other drugs or medical devices.
5. Active eye infection (including but not limited to: blepharitis, infectious conjunctivitis, keratitis, sclerotitis, endophthalmitis) in target eye or contralateral eye within 30 days prior to enrollment.
6. Ocular surface malignant tumor.
7. A history of allergic reaction or allergy to sodium luciferin, allergy to protein products used for treatment or diagnosis, allergy to ≥ 2 drugs or non-drug factors, or current allergic disease.
8. current in an infectious disease requiring oral, intramuscular or intravenous administration.
9. Patients with systemic immune diseases.
10. Any uncontrolled clinical problems (such as severe mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant neoplasms).
11. Not effective contraception.
12. In uncontrolled hypertension, systolic is no less than 160 mmhg, diastolic is no less than 100 mmhg.
13. In uncontrolled diabetes, fasting glucose is no less than 10.0umol/L.
14. Renal insufficiency, serum creatinine is more than 133umol/L.
15. Arrhythmia, myocardial ischemia, myocardial infarction (diagnosed by electrocardiogram).
16. Liver dysfunction, al ANINE aminotransferase and aspartate aminotransferase levels are higher than 80 IU/L.
17. Platelet level is below 100,000 /uL or above 450,000 /uL.
18. Hemoglobin level is below 10.0g/dL (male) or 9.0g/dL (female).
19. No anticoagulant was used, prothrombin time is higher than 16s, and thrombin time of activated part is higher than 50s.
20. HIV infection (HIV-positive).
21. Subjects lack compliance with the study or the ability to sign informed consent.
22. There are currently signs of systemic infection, including fever and ongoing antibiotic treatment (in this study, systemic infection was defined as deviation from normal values of white blood cells, lymphocytes, and neutrophils on routine blood tests).
23. Administration of Glucocorticoids and other systemic immunosuppressive drugs.
24. The investigator judges other conditions unsuitable for the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Effective clearance of HSV-1 genome | 12 months
  Judge HSV-1 genome clearance effective according to DNA sequencing results by methods of Plaque assay,Elisa,PCR etc.
Rate of reblindness in 3 participants with Refractory HSV Keratitis | 12 months
  180 days after corneal surgical, calculate rate of reblindness of treated eye in 3 participants.
HSV-1 virus testing outcome of the intervention eye | 12 months
  Herpes virus content before and after treatment were determinated by methods of plaque assay, ELISA, PCR etc. Compare the viral content changes with baseline.

SECONDARY OUTCOMES:
Corneal graft survival time | 12 months
  Observe the survival time of grafted cornea in participants, whether the grafted cornea is transparency or opacity.
Visual improvement compared with baseline | 12 months
  Judge the visual recovery progress according to visual examination results on day 3±1，7±2，30±7，90±14，180±21，360±31.
Concentration of dose limiting toxicities | 12 months
  Observe and record AE,SAE incidence of dose limiting toxicities related with BD111 administration.
Concentration of maximum tolerated dose | 12 months
  Observe and record AE,SAE at maximum tolerated dose when occurs dose limiting toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Yujia Cai, PhD, Principal Investigator — Shanghai BDgene Co., Ltd.
Locations (1):
- Eye & Ent Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei A, Yin D, Zhai Z, Ling S, Le H, Tian L, Xu J, Paludan SR, Cai Y, Hong J. In vivo CRISPR gene editing in patients with herpetic stromal keratitis. Mol Ther. 2023 Nov 1;31(11):3163-3175. doi: 10.1016/j.ymthe.2023.08.021. Epub 2023 Aug 31. PMID 37658603

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT04560790/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT04560790/ICF_000.pdf